CLINICAL TRIAL: NCT00775632
Title: A Phase II Randomized Study Comparing Low Dose Alemtuzumab and Cyclosporine With Standard of Care for the Prevention of Chronic Extensive GVHD for Patients Undergoing Allogeneic Peripheral Blood Stem Cell Transplantation (PBSCT) for Hematological Malignancies
Brief Title: Alemtuzumab and Cyclosporine for the Prevention of Graft vs Host Disease After Stem Cell Transplants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 07-0436C
Record Dates: First submitted 2008-10-16; First posted 2008-10-20 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Graft Versus Host Disease; Bone Marrow Transplantation
Keywords: Graft Versus Host Disease; Alemtuzumab; Campath; Bone Marrow Transplants
MeSH Terms: conditions — Graft vs Host Disease | interventions — Alemtuzumab; Mycophenolic Acid; Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator): The current standard of care for GVHD prophylaxis at Princess Margaret Hospital is cyclosporine and Mycophenolate or cyclosporine and methotrexate.
  Interventions: Drug: mycophenolate or cyclosporine and methotrexate
- Cyclosporine and Campath (Experimental): The efficacy of experimental arm will be tested against standard of care for prevention of Chronic extensive GVHD.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — A new GVHD prevention strategy will be tested against established GVHD prophylaxis in patients undergoing matched sibling donor transplant using peripheral blood stem cells.
  Arms: Cyclosporine and Campath
Drug: mycophenolate or cyclosporine and methotrexate — One of the two GVHD prophylaxis used at PMH-either cyclosporine and mycophenolate or cyclosporine and methotrexate
  Arms: Standard of Care

SUMMARY:
Graft versus host disease (GVHD) is one of the common complications after stem cell transplant. This is a complication, which happens when the new stem cells from the donor attack other cells in the body of the transplant recipient.

Recently, an antibody (protein) called alemtuzumab or Campath has been found to be effective in the prevention of Graft vs. Host Disease.

Previous studies have shown a low risk of GVHD with alemtuzumab, however the risk of disease recurrence was high. Previous studies have used a high dose of alemtuzumab. The purpose of this study is:

* To find if by lowering the dose of alemtuzumab, can serious GVHD be prevented without increasing the risk of relapse (your condition getting worse).
* To find whether low dose of alemtuzumab in combination with cyclosporine can prevent GVHD more effectively when compared to current standard of care and does not increase the risk of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a hematological malignancy
* Peripheral blood as source of stem cells
* Able to give informed consent
* Availability of 6/6 matched sibling donor
* Fit for transplant using a conventional or reduced intensity approach

Exclusion Criteria:

* AST/ALT >3 x IULN at the time of transplant
* Serum creatinine > 1.5 x IULN at the time of transplant
* Prior allogeneic transplant
* Syngeneic donor
* Active uncontrolled infection
* HIV positive
* Pregnancy at the time of BMT

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Chronic extensive GVHD at 1-year (yes vs. no) | 12 months from the date of transplant

CONTACTS AND LOCATIONS:
Overall Officials: Vikas Gupta, MD, Principal Investigator — University Heath Network
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada